CLINICAL TRIAL: NCT01756404
Title: A Double-Blind, Randomized, Placebo-Controlled, Sequential Cohort Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Multiple Ascending Oral Doses of JNJ-28431754 in Otherwise Healthy Obese Male and Female Subjects
Brief Title: Study to Assess the Pharmacokinetics, Pharmacodynamics, and Safety of Canagliflozin (JNJ-28431754) in Otherwise Healthy Obese Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: CR013765; 28431754NAP1008 (Other: Johnson & Johnson Pharmaceutical Research & Development, L.L.C.)
Record Dates: First submitted 2012-12-20; First posted 2012-12-25 (Estimated); Last update posted 2018-12-13 (Actual); Status verified 2018-12

CONDITIONS: Healthy
Keywords: Healthy; Canagliflozin (JNJ-28431754); Pharmacokinetics; Pharmacodynamics; Obesity
MeSH Terms: conditions — Obesity | interventions — Canagliflozin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

ARMS (5):
- Cohort 1 (Experimental): Each volunteer will receive a total daily dose of 30 mg of canagliflozin (JNJ-28431754) or placebo (inactive medication) on Days 1 through 14.
  Interventions: Drug: Canagliflozin (JNJ-28431754); Drug: Placebo
- Cohort 2 (Experimental): Each volunteer will receive a total daily dose of 100 mg of canagliflozin (JNJ-28431754) or placebo (inactive medication) on Days 1 through 14.
  Interventions: Drug: Canagliflozin (JNJ-28431754); Drug: Placebo
- Cohort 3 (Experimental): Each volunteer will receive a total daily dose of 300 mg of canagliflozin (JNJ-28431754) or placebo (inactive medication) on Days 1 through 14.
  Interventions: Drug: Canagliflozin (JNJ-28431754); Drug: Placebo
- Cohort 4 (Experimental): Each volunteer will receive a total daily dose of 600 mg of canagliflozin (JNJ-28431754) or placebo (inactive medication) on Days 1 through 14.
  Interventions: Drug: Canagliflozin (JNJ-28431754); Drug: Placebo
- Cohort 5 (Experimental): Each volunteer will receive 300 mg of canagliflozin (JNJ-28431754) twice daily (600 mg total daily dose) or placebo (inactive medication) twice daily on Days 1 through 14.
  Interventions: Drug: Canagliflozin (JNJ-28431754); Drug: Placebo

INTERVENTIONS:
Drug: Canagliflozin (JNJ-28431754) — A 30mg/day, 100 mg/day, 300 mg/day, or 600 mg/day liquid dose administered once daily; a 300mg/day liquid dose administered in 2 divided doses (2x150 mg); or a 600 mg/day liquid dose administered in 2 divided doses (2x300 mg) using an oral (by mouth) liquid dispenser on Days 1 through 14.
  Other Names: JNJ-28431754
Drug: Placebo — Matching placebo (inactive medication) liquid dose(s) administered using an oral liquid dispenser once or twice daily on Days 1 through 14.

SUMMARY:
The purpose of this study is to assess the pharmacokinetics (ie, how the body affects the drug) and pharmacodynamics (ie, how the drug affects the body) of increasing doses of canagliflozin (JNJ-28431754) in healthy obese volunteers.

DETAILED DESCRIPTION:
This study will be a single-center, randomized (the treatment is assigned by chance), double-blind (neither investigator nor volunteer knows the identity of the assigned treatment), placebo-controlled (one of the study medications is inactive), ascending multiple dose study (increasing doses of study medication) to assess the pharmacokinetics and pharmacodynamics of canagliflozin (a drug currently being investigated for the treatment of type 2 diabetes mellitus) in otherwise healthy obese volunteers. The study will consist of 3 phases: a screening phase, a double-blind treatment phase, and an end of study (or follow-up) phase. Volunteers will be assigned to 5 cohorts (groups) made up of 16 otherwise healthy obese men and women. Within each group, 12 volunteers will be given canagliflozin once or twice daily and 4 volunteers will be given placebo (inactive medication) once or twice daily for 14 days. The dose of canagliflozin will be different for each of the 5 groups and the second group will not begin treatment until at least 21 days after the first group start treatment. This 21-day gap will be applied to all subsequent groups. Each volunteer will participate in the study for approximately 58 days.

ELIGIBILITY:
Inclusion Criteria:

* Volunteers must have a body mass index (BMI = weight in kg/height in m2) of 30.0 to 39.9 kg/m2
* Volunteers must be non-diabetic as confirmed by fasting plasma glucose <126 mg/dL
* Volunteers must be non-smoker or non-tobacco users (not smoked cigarettes or used tobacco-containing products for 3 months prior to screening)

Exclusion Criteria:

* History of or currently active illness considered to be clinically significant by the Investigator or any other illness that the Investigator considers should exclude the patient from the study or that could interfere with the interpretation of the study results
* History of having taken anti-obesity medications (prescription or non-prescription) within 3 months of the screening visit, or anticipates a need to take any of these drugs during the course of the study
* History of gastric banding, gastric bypass or other gastric-reduction surgery
* History of eating disorder or recent significant changes in body weight due to dieting or nutritional treatment

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2007-06-14 (Actual); Primary Completion 2007-12-05 (Actual); Study Completion 2007-12-05 (Actual)

PRIMARY OUTCOMES:
Change from baseline in urine glucose excretion per day | Day -1 (Baseline) up to Day 17
  The change from baseline in urine excretion per day will be compared following escalating doses of canagliflozin (JNJ-28431754).
Change from baseline in urine glucose excretion per hour | Day -1 (Baseline) up to Day 17
  The change from baseline in urine excretion per hour will be compared following escalating doses of canagliflozin (JNJ-28431754).
Visual analog scale (VAS) scores related to hunger, satiety, fullness and prospective food consumption | Day -2 up to Day 17
  Visual analog scale (VAS) scores will be obtained from the VAS questionnaire. In the VAS questionnaire, volunteers mark a point on a line (drawn between 2 statements) to indicate how they feel about the statements. The statements about hunger are as follows: "I am not hungry at all" and "I have never been hungrier". Other statements relate to satiety (feeling satisfied), feeling full and prospective food consumption. Scores will be compared following escalating doses of canagliflozin (JNJ-28431754).
Change from baseline in mean 24-hour plasma glucose concentrations | Day -1 (Baseline) up to Day 16
  The change from baseline in mean 24-hour plasma glucose concentrations will be compared following escalating doses of canagliflozin (JNJ-28431754).

SECONDARY OUTCOMES:
Renal threshold for glucose excretion | Up to Day 17
  The point at which glucose starts to appear in the urine is known as the renal threshold. The way in which the renal threshold varies in relation to the dose of canagliflozin (JNJ-28431754) will be calculated.
Change from baseline in mean 24-hour plasma insulin concentrations | Day -1 (Baseline) up to Day 14
  The change from baseline in mean 24-hour plasma insulin concentrations will be compared following escalating doses of canagliflozin (JNJ-28431754).
Change from baseline in mean 24-hour plasma C-peptide concentrations | Day -1 (Baseline) up to Day 14
  The change from baseline in mean 24-hour plasma C-peptide concentrations will be compared following escalating doses of canagliflozin (JNJ-28431754).
Change from baseline in glucose excursions (after breakfast) | Day -1 (Baseline) up to Day 14
  Defined as the difference between the maximum glucose values observed during the 4-hour post-meal period minus the mean of the premeal measurements. Results will be compared following escalating doses of canagliflozin (JNJ-28431754).
Change from baseline in insulin excursions (after breakfast) | Day -1 (Baseline) up to Day 14
  Defined as the difference between the maximum insulin values observed during the 4-hour post-meal period minus the mean of the premeal measurements. Results will be compared following escalating doses of canagliflozin (JNJ-28431754).
Change from baseline in beta cell function | Day -1 (Baseline) up to Day 14
  Beta cell function will be calculated from the glucose, insulin, and C-peptide measurements taken post-breakfast on Day -1 up to Day 14. Results will be compared following escalating doses of canagliflozin (JNJ-28431754).

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.
Locations (1):
- Miramar, Florida, United States

REFERENCES:
- See also: A Double-Blind, Randomized, Placebo-Controlled, Sequential Cohort Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Multiple Ascending Oral Doses of JNJ-28431754 in Otherwise Healthy Obese Male and Female Subjects. — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217051&parentIdentifier=CR013765&attachmentIdentifier=98324aa4-364f-45ab-bbcf-0be725103e98&fileName=CR013765_CSR.pdf&versionIdentifier=